CLINICAL TRIAL: NCT04911400
Title: Effects of Class III Elastics on Stability of Orthopaedic Class III Correction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sydney Local Health District (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: X19-0365
Record Dates: First submitted 2021-05-09; First posted 2021-06-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Class III Malocclusion; Underbite
Keywords: Class III Malocclusion; Orthodontic retention
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper-lower clear plastic retainers + Class III elastics (Experimental): Upper-lower clear plastic retainers + Class III elastics
  Interventions: Other: Upper-lower clear plastic retainers + Class III elastics
- Upper-lower clear plastic retainers (Active Comparator): Upper-lower clear plastic retainers
  Interventions: Other: Upper-lower clear plastic retainers

INTERVENTIONS:
Other: Upper-lower clear plastic retainers + Class III elastics — Addition of Class III elastics to clear plastic retainers
  Arms: Upper-lower clear plastic retainers + Class III elastics
Other: Upper-lower clear plastic retainers — Upper-lower clear plastic retainers
  Arms: Upper-lower clear plastic retainers

SUMMARY:
The purpose of this study is to evaluate the effects of adding elastics to orthodontic retainers on the stability of class III correction and whether it reduces the need for jaw surgery.

DETAILED DESCRIPTION:
Over the years many types of appliances have been recommended for retaining Class III correction in growing children such as intermaxillary splints, class III activator, Frankel 3, Class III twin block, continued use of face-mask and chin-cup. However, currently none of these are in routine use and there is no evidence on the long term effectiveness of any retention protocol for class III correction.

One of the most commonly used retainers following orthodontic treatment is clear plastic retainers. There are no studies that investigated whether using class III elastics in combination with clear plastic retainers improves the stability of class III correction and reduces the need for later jaw surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that completed their orthodontic treatment for the management of their skeletal class III with upper jaw retrusion that was treated with Class III orthopaedic appliances, followed by full fixed appliances.
* No congenital anomalies or craniofacial syndromes
* No other orthodontic treatment
* No medical history that effects growth

Exclusion Criteria:

* Congenital anomalies or craniofacial syndromes
* Other orthodontic treatment
* Medical history that effects growth

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Difference in overjet of participants in the 2 study arms | 5 years
  Measurement of overjet

SECONDARY OUTCOMES:
Need for jaw surgery | 5 years
  Need for surgery assessed by a panel of orthodontists
Difference in upper jaw position | 5 years
  The difference in SNA angle measured on cephalometric radiographs between groups
Difference in lower jaw position | 5 years
  The difference in SNB angle measured on cephalometric radiographs between groups
Difference in upper-lower jaw relationship | 5 years
  The difference in ANB angle measured on cephalometric radiographs between groups
Difference in upper incisor angulation | 5 years
  The difference in upper incisor angle measured on cephalometric radiographs between groups
Difference in lower incisor angulation | 5 years
  The difference in lower incisor angle measured on cephalometric radiographs between groups
Compliance and ease of use of both retention regimens | 5 years
  Questionnaire on the frequency and ease of use of both retainer regimens will be used
Effect of elastics on alignment retention | 5 years
  Little's irregularity index will be used to compare both groups
Periodontal health, including recession around the incisors | 5 years
  Presence of gingival recession and prominence of lower incisors will be evaluated for both groups

CONTACTS AND LOCATIONS:
Overall Officials: Oyku Dalci, DDS, PhD, Principal Investigator — Sydney Local Health District, The University of Sydney
Locations (2):
- Australia (2):
  - Chatswood Orthodontics, Chatswood, New South Wales
  - Sydney Dental Hospital, Surry Hills, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Owens D, Watkinson S, Harrison JE, Turner S, Worthington HV. Orthodontic treatment for prominent lower front teeth (Class III malocclusion) in children. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD003451. doi: 10.1002/14651858.CD003451.pub3. PMID 38597341